CLINICAL TRIAL: NCT01847105
Title: Assessing Patient Comfort in Silicone Hydrogel Contact Lenses When Cleaned and Stored in Two Different Multi-Purpose Disinfecting Solutions
Brief Title: Assessing Patient Comfort With Two Different Multi-Purpose Disinfecting Solutions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hom, Milton M., OD, FAAO (Individual)
Collaborators: Abbott Medical Optics (Industry)
Responsible Party: Principal Investigator, Milton M. Hom, OD, FAAO., Optometrist, Hom, Milton M., OD, FAAO
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-GHS Comfort Study
Record Dates: First submitted 2013-04-24; First posted 2013-05-06 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Contact Lens Solution Toxicity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- RevitaLens (Experimental): AMO's RevitaLens contact lens solution
  Interventions: Other: RevitaLens; Other: OptiFree PureMoist

INTERVENTIONS:
Other: RevitaLens — Multi-purpose disinfecting solution
  Other Names: AMO's RevitaLens
Other: OptiFree PureMoist — Multi-purpose disinfecting solution
  Other Names: Alcon's OptiFree PureMoist MPS

SUMMARY:
Tolerability is compared between two Multi-purpose disinfecting solutions (MPDS).

DETAILED DESCRIPTION:
According to recent surveys of contact lens fitters, the most prescribed treatments for contact lens dryness are: more frequent replacement schedule (24%), refit into different material (23%), rewetting drops (21%) and change care system (15%). Changing care systems has been a standard treatment for CL discomfort for many years. In the same survey, 30% of practitioners felt there is absolutely no difference among solutions with respect to reducing dryness and discomfort.

The investigators set out to compare the clinical performance of these two solutions: AMO's RevitaLens and Alcon's Opti-Free PureMoist.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and over inclusive.
2. Males or females
3. Patient is in generally good & stable overall health.
4. Patient likely to comply with study guidelines & study visits.
5. Informed consent signed.
6. Are willing/able to return for all required study visits.
7. Are willing/able to follow instructions from the study investigator and his/her staff.
8. Have signed informed consent approved by Institutional Review Board or Independent Ethics Committee.

Exclusion Criteria:

1. Corneal refractive surgery within 6 months of this study.
2. Intra-ocular surgery within 6 months or ocular laser surgery within 6 months.
3. Ocular pathology (includes glaucoma and cataract), which could impact results and/or place patient at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Self-reported comfort scores with contact lens care systems | 14 days
  Comfort measured by questionnaires covering positive and negative attributes of contact lens wear

CONTACTS AND LOCATIONS:
Overall Officials: Milton M Hom, OD FAAO, Principal Investigator
Locations (3):
- United States (3):
  - Milton M. Hom, OD, FAAO, Azusa, California
  - Kirk L. Smick, OD, FAAO., Morrow, Georgia
  - Ian Ben Gaddie, OD, FAAO., Louisville, Kentucky